CLINICAL TRIAL: NCT00509899
Title: A Phase 1/2, Open-Label Study of the JAK2 Inhibitor INCB018424 Administered Orally to Patients With Primary Myelofibrosis (PMF) and Post Polycythemia Vera/Essential Thrombocythemia Myelofibrosis (Post-PV/ET)
Brief Title: Open Label Ruxolitinib (INCB018424) in Patients With Myelofibrosis and Post Polycythemia Vera/Essential Thrombocythemia Myelofibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-251
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Results first posted 2012-08-02 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Myelofibrosis; Polycythemia Vera; Thrombocytosis
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Thrombocytosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib (Experimental): All participants received oral ruxolitinib. Patients began treatment with either 10 mg twice a day (bid), 15 mg bid, 25 mg bid, 50 mg bid, 25 mg once a day (qd), 50 mg qd, 100 mg qd, or 200 mg qd, depending on the time period when they entered the study. The doses were titrated based on efficacy and safety to a maximum of 25 mg bid for patients who entered the study after sufficient dosing information had been obtained to define the maximum dose for patients in the study. Patients could continue receiving treatment indefinitely if receiving benefit at a dose that continues to maintain benefit but does not exceed a maximum dose of 25 mg BID.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — 5 and 25 mg tablets with a daily dosing range from 10 to 200 mg qd or bid.
  Other Names: INCB018424; Jakafi(TM)

SUMMARY:
To determine the safety, tolerability and effectiveness of ruxolitinib (INCB018424), administered orally to patients with Primary Myelofibrosis (PMF), Post Polycythemia Vera Myelofibrosis (PPV-MF) and Essential Thrombocythemia Myelofibrosis (PET-MF).

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, dose escalation study of ruxolitinib, a small molecule Janus kinase (JAK) inhibitor, administered orally to patients with PMF, PPEV-MF or PET-MF. The study is comprised of 3 parts:

Part 1: Dose escalation and determination of maximum tolerated dose (complete).

Part 2: Exploration of alternative dosing schedules (complete).

Part 3: Further evaluation of selected dose regimens, including additional response measures to explore effect of ruxolitinib on symptoms and other parameters including daily physical activity and long-term survival (ongoing).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PMF or Post-PV/ET MF
* Patients with myelofibrosis requiring therapy
* Adequate bone marrow reserve

Exclusion Criteria:

* Received anti-cancer medications or investigational therapy in the past 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center, Houston, TX; Ayalew Tefferi, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (2):
- United States (2):
  - Rochester, Minnesota
  - Houston, Texas

REFERENCES:
- [Result] Verstovsek S, Kantarjian H, Mesa RA, Pardanani AD, Cortes-Franco J, Thomas DA, Estrov Z, Fridman JS, Bradley EC, Erickson-Viitanen S, Vaddi K, Levy R, Tefferi A. Safety and efficacy of INCB018424, a JAK1 and JAK2 inhibitor, in myelofibrosis. N Engl J Med. 2010 Sep 16;363(12):1117-27. doi: 10.1056/NEJMoa1002028. PMID 20843246
- [Result] Verstovsek S, Kantarjian HM, Estrov Z, Cortes JE, Thomas DA, Kadia T, Pierce S, Jabbour E, Borthakur G, Rumi E, Pungolino E, Morra E, Caramazza D, Cazzola M, Passamonti F. Long-term outcomes of 107 patients with myelofibrosis receiving JAK1/JAK2 inhibitor ruxolitinib: survival advantage in comparison to matched historical controls. Blood. 2012 Aug 9;120(6):1202-9. doi: 10.1182/blood-2012-02-414631. Epub 2012 Jun 20. PMID 22718840
- [Derived] Kvasnicka HM, Thiele J, Bueso-Ramos CE, Sun W, Cortes J, Kantarjian HM, Verstovsek S. Long-term effects of ruxolitinib versus best available therapy on bone marrow fibrosis in patients with myelofibrosis. J Hematol Oncol. 2018 Mar 15;11(1):42. doi: 10.1186/s13045-018-0585-5. PMID 29544547

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a non-randomized dose-ranging study. Participants were enrolled into the currently available cohort based on the timeframe when they entered the study.
Groups:
- 10 mg Bid: Participants received an initial dose of Ruxolitinib 10 mg twice a day (bid). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy to a maximum of 25 mg bid.
- 15 mg Bid: Participants received an initial dose of Ruxolitinib 15 mg twice a day (bid). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy to a maximum of 25 mg bid.
- 25 mg Bid: Participants received an initial dose of Ruxolitinib 25 mg twice a day (bid). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy.
- 50 mg Bid: Participants received an initial dose of Ruxolitinib 50 mg twice a day (bid). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy.
- 25 mg qd: Participants received an initial dose of Ruxolitinib 25 mg once a day (qd). Participants could continue in the study on their prescribed regimen indefinitely with dose adjustments for safety and efficacy.
- 50 mg qd: Participants received an initial dose of Ruxolitinib 50 mg once a day (qd). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy.
- 100 mg qd: Participants received an initial dose of Ruxolitinib 100 mg once a day (qd). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy.
- 200 mg qd: Participants received an initial dose of Ruxolitinib 200 mg once a day (qd). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy.
Period: Overall Study
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | 50 mg Bid | 25 mg qd | 50 mg qd | 100 mg qd | 200 mg qd
Started | 30 | 35 | 47 | 5 | 6 | 22 | 6 | 3
Completed | 14 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).) | 26 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).) | 27 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).) | 1 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).) | 1 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).) | 12 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).) | 5 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).) | 2 (Represents patients still on study at the data cut-off for the interim analysis (31 December 2009).)
Not Completed | 16 | 9 | 20 | 4 | 5 | 10 | 1 | 1
Not completed — Progressive disease | 1 | 3 | 5 | 1 | 0 | 1 | 0 | 0
Not completed — Unacceptable Toxicity | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 3 | 0 | 3 | 2 | 0 | 0
Not completed — Physician Decision | 4 | 2 | 7 | 0 | 1 | 4 | 0 | 0
Not completed — Intercurrent Illness | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 2 | 3 | 0 | 1 | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | 50 mg Bid | 25 mg qd | 50 mg qd | 100 mg qd | 200 mg qd | Total
Number analyzed (Participants) | 30 | 35 | 47 | 5 | 6 | 22 | 6 | 3 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.29) | 63.8 (9.57) | 63.9 (9.06) | 63.0 (8.37) | 57.3 (9.89) | 66.3 (6.66) | 71.5 (6.89) | 72.3 (6.43) | 63.9 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 16 | 2 | 1 | 12 | 1 | 1 | 57
  Male | 18 | 23 | 31 | 3 | 5 | 10 | 5 | 2 | 97
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  White | 28 | 35 | 45 | 5 | 6 | 20 | 5 | 3 | 147
  Other | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Disease sub-type [Number; unit: Participants]
  Primary myelofibrosis | 12 | 19 | 23 | 3 | 5 | 14 | 5 | 0 | 81
  Post-polycythemia vera-myelofibrosis | 13 | 10 | 15 | 2 | 1 | 4 | 1 | 3 | 49
  Post-essential thrombocythemia-myelofibrosis | 5 | 6 | 9 | 0 | 0 | 4 | 0 | 0 | 24
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (3.8) | 25.3 (4.4) | 26.2 (5.9) | 24.8 (2.9) | 24.7 (2.9) | 25.3 (4.5) | 25.8 (6.3) | 26.3 (3.8) | 25.7 (4.7)
Palpable spleen length below the costal margin [Mean (Standard Deviation); unit: cm] | 19.11 (8.2) | 18.47 (5.7) | 17.13 (8.9) | 13.0 (10.1) | 19.58 (10.5) | 20.0 (7.3) | 20.67 (6.6) | 18.33 (3.5) | 18.37 (7.8)
JAK2 V617F mutation status [Number; unit: participants] — JAK2V617F is a mutation in the pseudokinase domain of Janus Kinase 2 (JAK2) (at amino acid 617, valine to phenylalanine) that results in constitutive activation of JAK2. Mutation status was determined using a validated assay on bone marrow as well as peripheral blood.
  participants
    Negative | 1 | 5 | 5 | 1 | 4 | 7 | 1 | 0 | 24
    Positive | 22 | 29 | 39 | 2 | 2 | 15 | 2 | 3 | 114
    Unknown | 7 | 1 | 3 | 2 | 0 | 0 | 3 | 0 | 16
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) performance status measures patients' functional status on the following scale: 0=Fully active, no restrictions 1=Restricted in physically strenuous activity but ambulatory, able to carry out light work; 2=Ambulatory and capable of all selfcare, unable to carry out any work activities; Up and about > 50% of waking hours; 3=Limited selfcare, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Totally confined to bed or chair; 5=Dead.
  participants
    0 | 7 | 0 | 9 | 2 | 1 | 5 | 1 | 0 | 25
    1 | 19 | 32 | 33 | 3 | 4 | 14 | 5 | 3 | 113
    2 | 4 | 3 | 5 | 0 | 1 | 3 | 0 | 0 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-Emergent AEs are events occurring after first drug administration or worsened from baseline.
  Treatment-Related AEs are those with a definite, probable, possible or missing causality.
  A serious AE is a medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is a medical event requiring intervention to prevent 1 of the above.
  A severe or life-threatening AE is based on intensity, according to National Cancer Institute-Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) v3.0.
Time Frame: From Baseline to the interim clinical cut-off date (31 December 2009). The median time on study was 14.8 months, with a range of 26 days to 29.7 months. As of March 1, 2011 the total exposure to ruxolitinib was 269 patient-years.
Population: Safety population included all patients who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- All QD: Participants received an initial dose of Ruxolitinib 25, 50, 100 or 200 mg once a day (qd). Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy. Since the numbers of patients in 3 of the qd treatment groups were small, the 4 qd doses were combined to allow meaningful comparisons against the bid treatment groups.
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | 50 mg Bid | All QD
Number analyzed (Participants) | 30 | 35 | 47 | 5 | 37
participants
  Any Treatment-Emergent Adverse Event | 30 | 35 | 47 | 5 | 37
  Treatment-Related Adverse Events | 21 | 22 | 41 | 4 | 29
  Serious Adverse Events | 8 | 17 | 21 | 2 | 23
  Severe or Life-threatening Adverse Events | 21 | 25 | 39 | 3 | 28
  Study Drug Interrupted Due to Adverse Events | 9 | 9 | 20 | 3 | 23
  Discontinued Study Drug Due to Adverse Events | 6 | 0 | 7 | 2 | 5
  Study Drug Reduced Due to Adverse Events | 8 | 12 | 26 | 1 | 11

2. Primary Outcome: Percentage of Participants With Clinical Improvement (CI) Over Time
Description: Clinical improvement was defined according to the International Working Group Myelofibrosis Research and Treatment criteria, and required 1 of the following:
  1. A ≥ 2 g/dL increase in Hemoglobin level or becoming transfusion independent;
  2. Either a ≥ 50% reduction in palpable splenomegaly if spleen was ≥ 10 cm at Baseline or a spleen palpable at > 5 cm at Baseline becomes not palpable;
  3. A ≥ 100% increase in platelet count and an absolute platelet count of ≥ 50,000 x 10^9/L or
  4. A ≥ 100% increase in absolute neutrophil count (ANC) and an ANC of ≥ 0.5 x 10^9/L.
Time Frame: Week 12, 24, 36, 48 and 60
Population: The intent-to-treat population included all patients who received at least 1 dose of study medication and had at least 1 follow-up assessment for safety and efficacy. N = the number of patients who had clinical response assessed during the time interval.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | 50 mg Bid | All QD
Number analyzed (Participants) | 25 | 34 | 42 | 5 | 32
percentage of participants
  12 Weeks [N=25, 34, 42, 5, 32] | 36.0 | 38.2 | 38.1 | 40.0 | 34.4
  24 Weeks [N=21, 31, 40, 4, 29] | 42.9 | 51.6 | 37.5 | 75.0 | 37.9
  36 Weeks [N=18, 30, 36, 4, 25] | 66.7 | 56.7 | 38.9 | 50.0 | 56.0
  48 Weeks [N=17, 28, 36, 3, 23] | 47.1 | 67.9 | 41.7 | 33.3 | 56.5
  60 Weeks [N=15, 21, 33, 2, 21] | 53.3 | 66.7 | 54.5 | 50.0 | 61.9

3. Secondary Outcome: Percentage of Participants Achieving ≥ 50% Reduction From Baseline in Spleen Palpation Length Over Time
Description: For each visit, patients who had a missing value at the visit, dropped out of the study due to any reasons prior to the visit or had non-palpable spleen at baseline and then became palpable at the time of the visit were all considered as having not achieved the ≥ 50% reduction in spleen palpation length.
Time Frame: Baseline and Weeks 4, 8, 12, 24, 36, 48 and 60
Population: Intent to treat population. A total of 16 patients had either a splenectomy prior to study entry, missing Baseline spleen values or had spleen lengths reported as 0 cm and were excluded.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | 50 mg Bid | All QD
Number analyzed (Participants) | 27 | 34 | 37 | 4 | 36
percentage of participants
  Week 4 [N=27, 34, 37, 4, 36] | 33.3 | 38.2 | 43.2 | 75.0 | 30.6
  Week 8 [N=27, 34, 37, 4, 36] | 29.6 | 50.0 | 43.2 | 75.0 | 30.6
  Week 12 [N=27, 34, 37, 4, 36] | 33.3 | 47.1 | 54.1 | 75.0 | 33.3
  Week 24 [N=26, 34, 37, 4, 36] | 34.6 | 52.9 | 48.6 | 50.0 | 36.1
  Week 36 [N=26, 34, 37, 4, 36] | 30.8 | 47.1 | 43.2 | 50.0 | 36.1
  Week 48 [N=26, 33, 37, 4, 36] | 23.1 | 54.5 | 40.5 | 25.0 | 27.8
  Week 60 [N=25, 27, 37, 4, 36] | 20.0 | 51.9 | 43.2 | 25.0 | 25.0

4. Secondary Outcome: Percentage of Participants With ≥ 35% Reduction From Baseline in Spleen Volume Over Time
Description: Spleen volume was assessed in a subgroup of 27 patients using magnetic resonance imaging (MRI) scans (or computed tomography (CT) scans in patients who were not candidates for MRI) of the abdomen in order to allow objective measurement of spleen volume using standard estimation techniques.
  For each visit, patients who had a missing value at the visit or dropped out of the study due to any reason prior to the visit were considered as not having achieved the ≥35% reduction in spleen volume.
Time Frame: Baseline, Weeks 4, 12, 24 and 48
Population: Patients with at least 1 Spleen-Volume Measurement. Patients who had not reached the visit were excluded from the analysis. In addition, at Week 48, 5 patients who did not have MRI measurement due to a protocol amendment were considered as not evaluable and were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Bid | 15 mg Bid
Number analyzed (Participants) | 2 | 25
percentage of participants
  Week 4 [N= 2, 25] | 0.0 | 44.0
  Week 12 [N= 2, 25] | 0.0 | 48.0
  Week 24 [N= 2, 25] | 0.0 | 44.0
  Week 48 [N= 2, 20] | 0.0 | 40.0

5. Secondary Outcome: Change From Baseline in Myelofibrosis Total Symptom Score at Week 24
Description: Symptoms of myelofibrosis were assessed using a modified Myelofibrosis Symptom Assessment Form (MFSAF). Abdominal discomfort, itching, muscle or bone pain, and night sweats are prominent and troubling symptoms in patients with MF. Therefore, the MFSAF-derived responses for these symptoms were analyzed as a total symptom score. Each symptom was assessed on a scale from 0 (absent), 1 (most favorable) to 10 (worst). The total symptom score is a sum of the individual scores and ranges from 0-40. A higher score indicates worse symptoms hence a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population for whom data was available. The MFSAF was implemented by protocol amendment while the study was ongoing. Hence data are available for only approximately 50% of enrolled patients. This analysis includes patients with a Baseline total symptom score ≥ 0; 8 patients were excluded because they had a Baseline score = 0.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | All QD
Number analyzed (Participants) | 9 | 26 | 11 | 17
scores on a scale | -4.7 (5.89) | -5.6 (7.82) | 0.9 (8.37) | -6.5 (6.38)

6. Secondary Outcome: Change From Baseline to Week 24 in Health-Related Quality of Life
Description: Health-related Quality of Life was assessed using the Global Health Status/Quality of Life Scale of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). This scale ranges from 0 to 100, with higher scores indicating higher quality of life.
Time Frame: Baseline and Week 24
Population: The safety population included all subjects who received at least 1 dose of study medication, and for whom data was available at both time points. The EORTC QLQ C30 was implemented by protocol amendment and as a result this data are available for only approximately 50% of the enrolled patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | All QD
Number analyzed (Participants) | 9 | 28 | 13 | 20
units on a scale | 14.81 (21.968) | 12.80 (22.620) | 0.63 (20.254) | 9.16 (28.725)

7. Secondary Outcome: Change From Baseline in Body Weight Over Time
Time Frame: Baseline and Weeks 4, 8, 12, 24, 36, 48 and 60.
Population: Intent-to-treat population for patients who had reached each time point and for whom data was available.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- All Participants: All participants received ruxolitinib at varying initial dose and regimen. Participants could continue in the study on their prescribed regimen indefinitely if receiving benefit with dose adjustments for safety and efficacy.
Arm/Group | All Participants
Number analyzed (Participants) | 146
kg
  Week 4 [n=139] | 0.30 (2.656)
  Week 8 [n=137] | 1.59 (2.773)
  Week 12 [n=129] | 2.44 (3.596)
  Week 24 [n=115] | 4.44 (4.422)
  Week 36 [n=104] | 5.58 (4.790)
  Week 48 [n=99] | 6.35 (5.845)
  Week 60 [n=83] | 6.60 (5.451)

8. Secondary Outcome: Change From Baseline to Week 24 in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG performance status measures patients' functional status on the following scale:
  * 0=Fully active, no restrictions;
  * 1=Restricted in physically strenuous activity but ambulatory, able to carry out light work;
  * 2=Ambulatory and capable of all selfcare, unable to carry out any work activities; Up and about > 50% of waking hours;
  * 3=Limited selfcare, confined to bed or chair more than 50% of waking hours;
  * 4=Completely disabled. Totally confined to bed or chair;
  * 5=Dead.
  Data reported indicate the number of participants with a change from Baseline score of -2, -1, 0 and 1.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population for patients who had reached each time point and for whom data was available.
Measure: Number; unit: participants
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | 50 mg Bid | All QD
Number analyzed (Participants) | 20 | 31 | 39 | 4 | 29
participants
  Change from Baseline of -2 | 1 | 0 | 1 | 0 | 0
  Change from Baseline of -1 | 4 | 15 | 16 | 2 | 15
  Change from Baseline of 0 | 12 | 16 | 18 | 1 | 11
  Change from Baseline of 1 | 3 | 0 | 4 | 1 | 3

ADVERSE EVENTS:
Arm/Group | 10 mg Bid | 15 mg Bid | 25 mg Bid | 50 mg Bid | All QD
Serious Adverse Events (participants affected / at risk) | 8/30 | 17/35 | 21/47 | 2/5 | 23/37
Other Adverse Events (participants affected / at risk) | 29/30 | 35/35 | 47/47 | 5/5 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Bid (N=30) | 15 mg Bid (N=35) | 25 mg Bid (N=47) | 50 mg Bid (N=5) | All QD (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 3 | 2 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 1
General symptom (General disorders) | 0 | 0 | 0 | 0 | 2
Hyperpyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 3 | 0 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 1 | 5
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Bid (N=30) | 15 mg Bid (N=35) | 25 mg Bid (N=47) | 50 mg Bid (N=5) | All QD (N=37)
Anaemia (Blood and lymphatic system disorders) | 14 | 14 | 27 | 0 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 11 | 29 | 4 | 14
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 2 | 1 | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 12 | 15 | 1 | 6
Nausea (Gastrointestinal disorders) | 7 | 4 | 6 | 1 | 6
Vomiting (Gastrointestinal disorders) | 4 | 4 | 6 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 6 | 5 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 4 | 4 | 1 | 3
Constipation (Gastrointestinal disorders) | 3 | 5 | 4 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 7 | 10 | 11 | 1 | 7
Edema peripheral (General disorders) | 2 | 8 | 10 | 3 | 0
Pyrexia (General disorders) | 1 | 4 | 6 | 2 | 5
Oedema (General disorders) | 2 | 1 | 5 | 0 | 0
Chills (General disorders) | 1 | 2 | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 4
Pitting oedema (General disorders) | 0 | 0 | 0 | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 1 | 1 | 3 | 1 | 3
Caput medusae (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 5 | 1 | 5
Pneumonia (Infections and infestations) | 0 | 3 | 4 | 0 | 6
Urinary tract infection (Infections and infestations) | 3 | 2 | 4 | 0 | 2
Bronchitis (Infections and infestations) | 2 | 3 | 3 | 0 | 2
Herpes zoster (Infections and infestations) | 4 | 0 | 5 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 4 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 4 | 0 | 4
Influenza (Infections and infestations) | 1 | 3 | 2 | 0 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 4 | 4 | 0 | 6
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 6 | 7 | 7 | 0 | 7
Weight increased (Investigations) | 3 | 4 | 9 | 1 | 8
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 4 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 0 | 3
Weight decreased (Investigations) | 2 | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 1 | 0 | 0
Arterial bruit (Investigations) | 0 | 0 | 0 | 1 | 1
Troponin increased (Investigations) | 0 | 2 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 7 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 11 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8 | 5 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4 | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 1
Dysplastic naevus syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 6 | 5 | 3 | 6
Dizziness (Nervous system disorders) | 2 | 3 | 3 | 0 | 5
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 2 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 4 | 3 | 0 | 6
Depression (Psychiatric disorders) | 2 | 1 | 4 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 3 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 3 | 2 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 3 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 9 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 7 | 0 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 5 | 9 | 0 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 6 | 5 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 6 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 0 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Haematoma (Vascular disorders) | 1 | 3 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study; provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.